CLINICAL TRIAL: NCT01046539
Title: A Phase 1 Study to Evaluate the Pharmacodynamics of RDC-0313 Coadministered With Buprenorphine to Opioid-Experienced Healthy Adults
Brief Title: Phase 1 Study to Evaluate RDC-0313 Coadministered With Buprenorphine to Opioid-Experienced Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Reese Jones, M.D. / Principal Investigator, Langley Porter Psychiatric Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK33-008
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2010-07

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — ALKS-33; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RDC-0313 + Buprenorphine (Active Comparator): Cohort 1 (1 and 4 mg) + 8 mg Cohort 2 (dependent on Cohort 1 results)
  Interventions: Drug: RDC-0313 + Buprenorphine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDC-0313 + Buprenorphine — 1 and 4 mg (1 dose for each) + 8 mg
  Arms: RDC-0313 + Buprenorphine
Drug: Placebo — 0 mg
  Arms: Placebo

SUMMARY:
This is a single site, double-blind, randomized, placebo-controlled, crossover study to assess the pharmacodynamics (PD) of RDC-0313 coadministered with buprenorphine in 12 healthy, opioid-experienced, non-treatment-seeking subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be capable of understanding and complying with the protocol and has signed the informed consent
* Must be 18-55 years of age
* Must have a body mass index of 18.0-30.0 kg/m2 at screening
* Female subjects must agree to use an acceptable method of contraception from date of consent and until two weeks after the last dose
* Subjects must be willing not to use alcohol-, tobacco, caffeine-, or xanthine-containing products while resident at inpatient facility
* Subjects must be an experienced opioid user who meets the following criteria: 1) has used opioids for non-therapeutic purposes (ie, for psychoactive effects) on at least 10 occasions in the past five years; 2) has used opioids at least 2 times in the two years prior to screening; and 3) is not physically dependent on opioids, as assessed by medical history and naloxone challenge performed at screening

Exclusion Criteria:

* Must not have any current or piror significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders.
* Must not have current or past opioid, alcohol, or other durg dependence (excluding nicotine and caffeine) or showing signs of withdrawal following the naloxone (Narcan) challenge.
* Please contact site for additional information about other exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics (PD) of study drug | 24 hour period
VAS Scores | 24 Hours period
Pupuillometry Assessments | 24 Hour Period
Subjective Symptoms | 15 min pre and post nal, 3 hrs post bup admin

SECONDARY OUTCOMES:
To determine pharmacokinetics (PK) and evaluate safety and tolerability of study drug | 24 hour period
Max plasma concentration | 24 Hour Period
Time to maximum plasma concentration | 24 Hour Period
Area under the concentration time curve (AUC) | 24 Hour Period
Additional PK parameters may be analyzed | As appropriate

CONTACTS AND LOCATIONS:
Locations (1):
- Langley Porter Psychiatric Hospital, San Francisco, California, United States